CLINICAL TRIAL: NCT05107388
Title: AAREN: Continuous Glucose Monitoring Profile Description Under Alpelisib treAtment in Patients With Advanced bREast Cancer
Brief Title: Continuous Glucose Monitoring Profile Description Under Alpelisib treAtment in Patients With Advanced bREast Cancer
Acronym: AAREN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/609
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Diabetes
Keywords: Breast Cancer, Alpelisib, hyperglycemia
MeSH Terms: conditions — Breast Neoplasms; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous interstitial glucose measurements (Experimental): Variations of interstitial glucose are measured during 14 days with FreeStyle Libre Pro
  Interventions: Device: FreeStyle Libre Pro

INTERVENTIONS:
Device: FreeStyle Libre Pro — Measurements of interstitial glucose variations with FreeStyle Libre Pro

SUMMARY:
The purpose of this study is to describe the glycemic profile of postmenopausal women treated with alpelisib plus fulvestrant using a continuous blood sugar monitoring device (FreeStyle Libre Pro) over 14 days

DETAILED DESCRIPTION:
AAREN is a monocentric prospective study monitoring glycemic profile in patients treated with alpelisib plus fulvestrant. Patients will wear a noninvasive glucose monitoring sensor, the Freestyle Libre Pro for a 14 day period. Forty patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Women suffering breast cancer and eligible to treatment with Alpelisib
2. Age ≥18 years
3. Menopausal women (for at least 24 months)
4. Informed Consent Form signed

Exclusion Criteria:

1. Men
2. Pregnant ou child-bearing potential women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of hyperglycemia | Day 14
  In percentage, measured before breakfast and diner (fasting blood glucose).
  Hyperglycemia defined as follows:
  * if diabetes de novo:
    * capillar or interstitial fasting blood glucose ≥ 1,50 g/L,
    * OR postprandial interstitial glucose ≥ 2 g/L
    * OR glucose monitoring indicator ≥ 6,5%
  * if worsening pre-existing diabetes:
    * increased capillar or interstitial fasting blood glucose ≥ 0,50 g/L compared to average fasting blood glucose at J-3, J-2 and J-1
    * AND postprandial interstitial glucose ≥ + 1,00 g/L compared to average fasting blood glucose at J-3, J-2 et J-1 OR average blood glucose ≥ +0,50 g/L

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BOROT, MD, PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No